CLINICAL TRIAL: NCT03229837
Title: Pediatric Patient-Reported Outcomes (PEPR) for Childhood Cancer Survivors: Clinical Validity Study
Brief Title: Validation Study of Pediatric Patient-Reported Outcomes
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: PEPR II; U19AR069525 (NIH)
Record Dates: First submitted 2017-07-07; First posted 2017-07-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Tumor; Malignancy
Keywords: Construct validity; Minimally important differences; Patient-reported outcomes; Pediatric cancer survivors; PROMIS pediatric measures
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Survivors of childhood cancer often suffer treatment-related toxicities, including chronic health conditions, high symptom burden and emotional distress, and decremented functional status and quality of life. Although some patient-reported outcome (PRO) tools are available for survivors of childhood cancer younger than 18 years old, very few studies have been designed to evaluate longitudinal measurement properties of these PRO tools. In this study the investigators propose to recruit participants from a cohort of diverse childhood cancer survivors who were treated at St. Jude Children's Research Hospital (St. Jude) to improve assessment tools for PROs and health-related quality of life (HRQOL).

The purpose of this study is to measure the link between Patient Reported Outcome Measurement Information System (PROMIS) and clinical assessments of childhood cancer survivors over time. PROMIS is a questionnaire that measures patient-reported outcomes in adults and children.

The study plans to enroll 300 children. Surveys will be completed by the children and their parents/legal guardians (a total of 600 surveys).

PRIMARY OBJECTIVES:

1. To evaluate the longitudinal construct validity of the PROMIS Pediatric measures for childhood cancer survivors by testing the association of change in PROMIS PRO scores and the change in health status measured by objective clinical assessment. Age at baseline and sex will be included in the analysis.
2. To establish clinically meaningful classifications of the PROMIS Pediatric measures for childhood cancer survivors by referring PROMIS PRO scores to health status measured by clinical assessment. Age at baseline and sex will be included in the analysis.
3. To estimate the minimally important differences (MIDs) of the PROMIS Pediatric measures by referring to the change of health status evaluated by anchor-based anchors and patient-based anchors for childhood cancer survivors. Age at baseline and sex will be included in the analysis.

DETAILED DESCRIPTION:
A longitudinal framework was designed to collect data from childhood cancer survivors (8-18.9 years of age) and parents of participating cancer survivors (i.e., dyads) when they visit the After Completion of Therapy (ACT) clinic at St. Jude in three consecutive years (approximately 1 year apart; T1, T2, and T3).

Participants will complete pediatric patient-reported outcomes (PRO) survey/questionnaires, a neurocognitive assessment and physical performance evaluation will be completed, and parental surveys will be conducted. In addition, any data collected as part of the SJLIFE protocol may also be used as part of this study.

1. The Pediatric PRO survey/questionnaires collection information on PROs. They include questions about general health, pain interference, fatigue, psychological stress experiences, stigma, sleep disturbance, sleep-related impairment, positive affect, meaning and purpose, depressive symptoms, anxiety, and physical function-mobility. Each cancer survivor will complete these during annual follow-up visits at three time points: years 1, 2 and 3. This process takes approximately 30-40 minutes.
2. Neurocognitive evaluation is done by tests given by a licensed or certified psychological examiner to evaluate how the participant processes information. The tests evaluate how problems are solved, how well information is remembered, how well the participant pays attention, how quickly they understand information, and their assessment of quality of life. The tests are commonly used standardized tests that take about 2 hours to complete.
3. Physical performance evaluation will measure heart and lung fitness, flexibility, mobility, muscle strength, endurance, balance and physical mobility. Testing takes about 2 hours to complete and includes six-minute walk test, walking speed test, muscle strength and flexibility, and balance.
4. The parental survey is a parent-report form (PRF) to be completed by parents/legal guardians of participants. Information collected on the PRF includes demographic information, parental quality of life, social support, family dynamics, parenting behaviors, and the child's health care utilization data. The child and parent data will be compared. Parental questionnaires will be completed at one time point, year 1, 2, or 3, and will take approximately 40 minutes to complete.

ELIGIBILITY:
Inclusion Criteria for Childhood Survivors:

* St. Jude childhood cancer survivors who have consented to SJLIFE;
* Age at assessment: 8-18.9 years at T1 (toward 20.9 years at T3);
* 2 years off therapy and > 5 years since diagnosis; and
* Agrees to complete three annual assessments during routinely scheduled ACT clinic appointments.

Exclusion Criteria for Childhood Survivors:

* Cancer-related or unrelated (e.g., genetic disorders) neurocognitive injuries that requires parents/proxies to complete the survey [e.g. intelligence quotient (IQ) <70];
* Inability to read and speak English; or
* Parent doesn't agree to participate in the parent part of the study.

Inclusion Criteria for Parents/Legal Guardians:

* Parent/legal guardian of St. Jude childhood cancer survivor aged 8-18.9 who is eligible to participate and has agreed to do so;
* Participant is not developmentally delayed, intellectually disabled or non-communicative; and
* Participant speaks and understands the English language.

Exclusion Criteria for Parents/Legal Guardians:

* Developmentally delayed, intellectually disabled or non-communicative;
* Unable to speak or understand the English language; and
* Child doesn't agree to participate in child part of the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from a cohort of diverse childhood cancer survivors who were treatment at St. Jude and their parents/legal guardians.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change of PROs | From baseline through 3 years
  The change of patient-reported outcome (PRO) between time points will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: I-Chan Huang, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols